CLINICAL TRIAL: NCT06036784
Title: A Phase 1 Single and Multiple Ascending Dose and Drug Drug Interaction Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of MBX 1416 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MBX Biosciences (Industry)
Collaborators: ProSciento, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: MBX-1P2001
Record Dates: First submitted 2023-08-28; First posted 2023-09-14 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Postbariatric Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MBX 1416 (Part A) (Experimental): Single ascending subcutaneous (SC) doses
  Interventions: Drug: MBX 1416 (Part A)
- MBX 1416 (Part B) (Experimental): Repeated ascending subcutaneous (SC) doses
  Interventions: Drug: MBX 1416 (Part B)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MBX 1416 (Part C) (Experimental): Single subcutaneous (SC) dose of MBX 1416, single dose of rosuvastatin and acetaminophen.
  Interventions: Drug: MBX 1416 (Part C)

INTERVENTIONS:
Drug: MBX 1416 (Part A) — Single Ascending subcutaneous (SC) dose of MBX 1416: 10mg, 30mg,100mg, 200mg
  Arms: MBX 1416 (Part A)
Drug: MBX 1416 (Part B) — Repeated ascending subcutaneous (SC) doses of MBX 1416: 10mg, 30mg, 100mg
  Arms: MBX 1416 (Part B)
Drug: Placebo — Single dose or repeated subcutaneous (SC) dose of placebo.
  Arms: Placebo
Drug: MBX 1416 (Part C) — Single subcutaneous (SC) dose of MBX 1416 and the single dose of rosuvastatin and acetaminophen pharmacokinetics. The doses selected for MBX 1416 in Part C will not exceed a dose of 200mg.
  Arms: MBX 1416 (Part C)

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple doses and Drug Drug Interaction of MBX 1416 in healthy volunteers

This study includes 3 parts. Part A involves a single dose of MBX 1416 or placebo taken as a subcutaneous injection (SC). Part B involves repeat doses of MBX 1416 or placebo taken as a subcutaneous injection (SC). Part C involves the evaluation of rosuvastatin and acetaminophen pharmacokinetics in the presence and absence of MBX 1416.

ELIGIBILITY:
Part A/B/C Inclusion Criteria:

1. Female and male adults, ages ≥ 18 and ≤ 65 years with a body mass index (BMI) ≥ 18 kg/m² to ≤ 30.0 kg/m² and fasting glucose < 100 mg/dL and HbA1c < 5.7%.
2. Female subjects of childbearing potential (WOCBP) and male subjects must use highly effective contraception.

Part A/B/C Exclusion Criteria:

1. Pregnant, lactating or intending to become pregnant during the study.
2. Use of weight-lowering pharmacotherapy or participation in a clinical weight control study within the previous 3 months prior to the first dose of study drug.
3. Presence of clinically significant ECG findings
4. Subjects with a prior history of any serious adverse reaction, hypersensitivity or angioedema to GLP-1 receptor agonists, study drug or drug components.
5. Abnormal laboratory results at Screening.
6. History of renal disease or abnormal kidney function tests at Screening
7. Presence of any clinically significant physical exam, ECG, or laboratory findings at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), Serious Adverse Events (SAEs) | Baseline through Day 29 (Part A) or Day 45 (Part B) and Day 21 (Part C)
Maximum Plasma Concentration (Cmax) | Baseline through Day 29 (Part A) or Day 45 (Part B) and Day 21 (Part C)

CONTACTS AND LOCATIONS:
Locations (1):
- MBX Biosciences Investigational Site, Chula Vista, California, United States

REFERENCES:
- [Derived] Fabbrini E, Koshkina A, Hackett M, Zhao M, Thalluri K, Hompesch M, Macias A, Schneider K, D'Alessio DA, DiMarchi RD, Azoulay S. Sustained Action of Imapextide, a Glucagon-Like Peptide-1 Receptor Antagonist, in Healthy Volunteers. J Clin Endocrinol Metab. 2025 Dec 24:dgaf691. doi: 10.1210/clinem/dgaf691. Online ahead of print. PMID 41437319